CLINICAL TRIAL: NCT02070367
Title: Somatosensory Assessment and Rehabilitation of Allodynia: the SARA Pilot Study
Brief Title: Somatosensory Assessment and Rehabilitation of Allodynia (SARA)
Acronym: SARA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-798
Record Dates: First submitted 2014-02-03; First posted 2014-02-25 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Complex Regional Pain Syndrome; Peripheral Nerve Injuries; Hand Fractures
Keywords: allodynia; complex regional pain syndrome; peripheral nerve injuries; clinical measurement properties
MeSH Terms: conditions — Complex Regional Pain Syndromes; Peripheral Nerve Injuries; Hyperalgesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Somatosensory rehabilitation (Experimental): Weekly sessions with a certified (RSDC) somatosensory therapist using distal vibro-tactile counter-stimulation to anatomically related territories of the area of allodynia. Participants will also be provided with a structured home exercise program.
  Interventions: Other: Somatosensory rehabilitation; Other: Usual treatment: physiotherapy
- Usual treatment (Active Comparator): Treatment as usual for condition Physiotherapy sessions
  Interventions: Other: Usual treatment: physiotherapy

INTERVENTIONS:
Other: Somatosensory rehabilitation
  Arms: Somatosensory rehabilitation
Other: Usual treatment: physiotherapy

SUMMARY:
This pilot study will test a new therapy, somatosensory rehabilitation, for the painful sensitivity experienced by persons with nerve injuries and/or complex regional pain syndrome (CRPS). Several methods for measuring pain and sensitivity that emphasize the person's evaluation of their own symptoms and the impact of these symptoms on their daily activities will also be tested to make sure they are consistent and accurate.

Previous research has suggested one of the assessments may also be used to assist in the identification of CRPS: this simple test will be evaluated to see if it can accurately identify persons with this disorder (for which there is currently no diagnostic test). Together, this will improve treatment of CRPS through early, accurate diagnosis and the ability to measure important changes in this painful condition, and set up future studies for this new rehabilitation treatment method.

DETAILED DESCRIPTION:
We will test four groups: persons with CRPS of one upper extremity, persons with recent hand fractures (<12 weeks) or peripheral nerve injuries with residual sensory deficits at the time of the study, and healthy normal volunteers with a battery of assessments for CRPS, including a technique to precisely localize and quantify static mechanical allodynia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a) Complex Regional Pain Syndrome or b) Peripheral Nerve Injury or c) recent hand trauma without peripheral nerve injury in a single upper extremity confirmed by physician or medical record.
* Participant and most responsible physician give consent to exclusive focus on somatosensory rehabilitation for the duration of the trial (6 months). The participant may continue any oral medications but any planned use of topical medication, injections or IV medication in the affected limb is contra-indicated. Use of these modalities in an emergency situation would of course take priority.

Exclusion Criteria:

* History of cardiac or vascular disease or known sensitivity to sympathetic stress or cold intolerance or medically unstable
* Confounding diagnoses: whiplash, nerve root compression, metabolic diseases such as diabetes or thyroid problems, and/or peripheral neuropathy
* Open wounds on testing sites
* Unable to provide informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-10; Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
McGill Pain Questionnaire | baseline to 6 month follow-up
  total number and intensity of sensory and affective pain descriptors selected by participant

SECONDARY OUTCOMES:
Pain subscale of the Patient-Rated Wrist and Hand Evaluation | Baseline to six months
  5 questions rating self-reported pain at rest, with movement, pain with lifting, worst pain and pain frequency.
Hamilton Inventory for Complex Regional Pain Syndrome | Baseline to 6 months
  Includes a both a patient-reported scale addressing symptoms, daily function and psychosocial concerns; and a clinician-based assessment of clinical signs
Radboud Evaluation of Sensitivity- English version | Baseline to 6 months
  self-reported evaluation of sensitivity in an area of injury/trauma

OTHER OUTCOMES:
10 test | Baseline to 3 months
  quick form of quantitative sensory testing for light touch sensation and hypersensitivity
Pain Catastrophizing Scale | Baseline to 6 months
  Measures pain-related beliefs
Allodynography | Baseline to 3 months
  a graphical technique to anatomically map allodynia associated with a specific nerve branch and assess the area and associated pressure threshold
Infra-red skin temperature measurement asymmetry | Baseline and 3 months
  Infra-red measures of skin temperature are taken over 3 specific areas (corresponding to the most distal autonomous innervation from the 3 major peripheral nerves of the upper limb) and symmetry is compared between the right and left arms. This measurement procedure is then repeated after a 30 second immersion of the right foot in ice water (5 degrees C).
Goniometric measurement of active range of motion (ROM) of the upper extremities | Baseline to 3 months
  Measures of affected and unaffected limbs (shoulder flexion and abduction, elbow flexion/extension, wrist flexion/extension, forearm pronation/supination, active functional ROM of the fingers, thumb opposition).
Dynamometry for grip and pinch strength | Baseline to 3 months
  bilateral measures of hand grip and pinch strength

CONTACTS AND LOCATIONS:
Overall Officials: Joy C MacDermid, PhD, Principal Investigator — School of Rehabilitation Sciences, McMaster University
Locations (1):
- Hamilton Health Science, General Site, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Packham TL, Fok D, Frederiksen K, Thabane L, Buckley N. Reliability of infrared thermometric measurements of skin temperature in the hand. J Hand Ther. 2012 Oct-Dec;25(4):358-61; quiz 362. doi: 10.1016/j.jht.2012.06.003. Epub 2012 Sep 10. PMID 22975739
- [Background] Packham T, MacDermid JC, Henry J, Bain JR. The Hamilton Inventory for Complex Regional Pain Syndrome: a cognitive debriefing study of the clinician-based component. J Hand Ther. 2012 Jan-Mar;25(1):97-111; quiz 112. doi: 10.1016/j.jht.2011.09.007. PMID 22265445
- [Derived] Packham T, MacDermid J, Bain J, Buckley N. Identification of complex regional pain syndrome in the upper limb: Skin temperature asymmetry after cold pressor test. Can J Pain. 2018 Aug 21;2(1):248-257. doi: 10.1080/24740527.2018.1504283. eCollection 2018. PMID 35005383
- [Derived] Packham TL, Spicher CJ, MacDermid JC, Quintal I, Buckley N. Evaluating a sensitive issue: reliability of a clinical evaluation for allodynia severity. Somatosens Mot Res. 2020 Mar;37(1):22-27. doi: 10.1080/08990220.2019.1704242. Epub 2019 Dec 20. PMID 31858880
- [Derived] Packham TL, Spicher CJ, MacDermid JC, Buckley ND. Allodynography: Reliability of a New Procedure for Objective Clinical Examination of Static Mechanical Allodynia. Pain Med. 2020 Jan 1;21(1):101-108. doi: 10.1093/pm/pnz045. PMID 30908579